CLINICAL TRIAL: NCT03357406
Title: Immediate Loading After Conventional and Ultrasonic Implant Site Preparation: a Multicenter Randomized Controlled Clinical Trial
Brief Title: Conventional and Ultrasonic Implant Site Preparation
Acronym: PI-DRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of International Piezosurgery Academy, International Piezosurgery Academy
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: piezo-drills
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Bone Atrophy, Alveolar
Keywords: implant; piezoelectric; drills; immediate loading
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Investigator, Outcomes Assessor
Masking Description: treatment method is masked till the surgical procedure, during which, both surgeon and patient are informed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edentulism side 1 (Experimental): ultrasound implant site preparation
  Interventions: Procedure: ultrasound implant site preparation
- edentulism side 2 (Active Comparator): conventional implant site preparation
  Interventions: Procedure: conventional implant site preparation

INTERVENTIONS:
Procedure: ultrasound implant site preparation — piezoelectric bone surgery will be used to create implant bone ostectomy
  Arms: edentulism side 1
Procedure: conventional implant site preparation — twist drills will be used to create implant bone ostectomy
  Arms: edentulism side 2

SUMMARY:
multi center study with randomized controlled trial design, split mouth

DETAILED DESCRIPTION:
The present study has been designed as a multicenter prospective randomized controlled trial design. Fifteen clinical centers will treat patients by inserting and immediately loading implants with two different surgical protocols. Each patient will receive two identical implants: after randomization, the test site will be prepared by ultrasonic microvibrations and the control site using twist drills. Both implants will be loaded with a provisional crown within 48 hours after surgery. For each inserted implant, collection of experimental parameters will be required up to 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

indications for two implant-supported single crowns with immediate loading in the upper or lower arch (in the incisor, canine or premolar area), based on accurate diagnosis and treatment planning; 2) implants can be in the same or in different quadrants; 3) implant sites must be performed in similar bone quality (i.e. both maxillary or mandibular); 4) the bone crest must be healed (at least three months elapsed after tooth loss); 5) presence of a residual bone crest with an adequate volume to allow the insertion of a 3.8x11.5 mm implant without any kind of regenerative procedure; 6) age of the patient >18 years; 7) patient willing and fully capable to comply with the study protocol; 8) written informed consent given;

Exclusion Criteria:

1. acute myocardial infarction within the past 2 months;
2. uncontrolled coagulation disorders;
3. uncontrolled diabetes (HBA1c > 7.5%);
4. radiotherapy to the head/neck district within the past 24 months;
5. immunocompromised patient (HIV infection or chemotherapy within the past 5 years);
6. present or past treatment with intravenous bisphosphonates;
7. psychological or psychiatric problems;
8. alcohol or drugs abuse Local exclusion criterion is the presence of uncontrolled or untreated periodontal disease (full mouth plaque score and full mouth bleeding score > 25%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
implant survival rate | two years after surgery
  how many implant are present in mouth

SECONDARY OUTCOMES:
implant success rate | two years after surgery
  implant stable and fulfilling success criteria
biomechanical complications | two years after surgery
  every complication linked to the crown, implant abutment structure
marginal bone loss | two years after surgery
  radiographically assessed bone level

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Director — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vercellotti T, Stacchi C, Russo C, Rebaudi A, Vincenzi G, Pratella U, Baldi D, Mozzati M, Monagheddu C, Sentineri R, Cuneo T, Di Alberti L, Carossa S, Schierano G. Ultrasonic implant site preparation using piezosurgery: a multicenter case series study analyzing 3,579 implants with a 1- to 3-year follow-up. Int J Periodontics Restorative Dent. 2014 Jan-Feb;34(1):11-8. doi: 10.11607/prd.1860. PMID 24396835
- [Background] Esposito M, Grusovin MG, Achille H, Coulthard P, Worthington HV. Interventions for replacing missing teeth: different times for loading dental implants. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD003878. doi: 10.1002/14651858.CD003878.pub4. PMID 19160225
- [Background] Khayat PG, Arnal HM, Tourbah BI, Sennerby L. Clinical outcome of dental implants placed with high insertion torques (up to 176 Ncm). Clin Implant Dent Relat Res. 2013 Apr;15(2):227-33. doi: 10.1111/j.1708-8208.2011.00351.x. Epub 2011 May 20. PMID 21599832